CLINICAL TRIAL: NCT02514200
Title: Treatment of Keratoconus With Advanced Corneal Crosslinking-II
Brief Title: Treatment of Keratoconus With Advanced CXL-II
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Umeå University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KXL2
Record Dates: First submitted 2015-07-30; First posted 2015-08-03 (Estimated); Last update posted 2018-05-16 (Actual); Status verified 2017-12

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus | interventions — Riboflavin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Topography-based CXL (KXL2) (Experimental): Individualized pulsed topography-based corneal crosslinking; 1 second on, 1 second off; 7.2J/cm2 - 15.0J/cm2; arcuate treatment zone. The Avedro KXL II™ System is used for the crosslinking after epithelial debridement in topical anesthesia and application of topical riboflavin every 3 minutes for 10 minutes.
  Interventions: Procedure: Topography-based CXL (KXL2); Drug: Riboflavin; Device: Avedro KXL II
- Conventional pulsed CXL (pCXL) (Active Comparator): Conventional pulsed corneal crosslinking; 1 second on, 1 second off; 5.4 J/cm2; 8 mm central treatment zone. The Avedro KXL II™ System is used for the crosslinking after epithelial debridement in topical anesthesia and application of topical riboflavin every 3 minutes for 10 minutes.
  Interventions: Procedure: Conventional pulsed CXL (pCXL); Drug: Riboflavin; Device: Avedro KXL II

INTERVENTIONS:
Procedure: Topography-based CXL (KXL2) — The keratoconus cornea is treated with epithelial debridement in local anesthesia, and then soaked in Riboflavin by repeated topical application every 3 minutes during 10 minutes. The cornea is then irradiated with pulsed ultraviolet light (1s on/1s off) in a topography-based arcuate shape with the Avedro KXL2® with an energy from 7.2-15.0 J/cm2 depending on the severity of the keratoconus.
  Arms: Topography-based CXL (KXL2)
Procedure: Conventional pulsed CXL (pCXL) — The keratoconus cornea is treated with epithelial debridement in local anesthesia, and then soaked in Riboflavin by repeated topical application every 3 minutes during 10 minutes. The cornea is then irradiated with pulsed ultraviolet light (1s on/1s off) in a central round 8mm zone with the Avedro KXL2® with an energy of 5.4 J/cm2.
  Arms: Conventional pulsed CXL (pCXL)
Drug: Riboflavin — Riboflavin is added topically immediately before the treatment every 3 minutes during 10 minutes in the eye to be treated
Device: Avedro KXL II — The KXL II™ System crosslinking device from Avedro, Inc. is used for ultraviolet irradiation of the cornea after riboflavin application in both treatment arms.

SUMMARY:
The purpose of this study is to determine whether individualized, topography-based corneal crosslinking for keratoconus can improve the optical outcomes of the treatment.

DETAILED DESCRIPTION:
The study is designed as a prospective, open label, randomized controlled trial involving patients aged 12 years or older of both genders with uni- or bilateral keratoconus planned for routine corneal crosslinking (CXL) at the Department of Clinical Sciences / Ophthalmology, Umeå University Hospital, Umeå, Sweden. The study involves 25+25 eyes with keratoconus, which are randomized to receive either conventional pulsed crosslinking with a uniform, universal 8 mm treatment pattern of 5.4 J/cm2 (pCXL; n=25), or a modified treatment - individualized topography-based corneal crosslinking (KXL2; n=25). In the latter treatment zone has an individualized arcuate shape and spares a 2 mm central optical zone. The size of the treatment zone is based on Pentacam HR® corneal tomography, and is determined by the transition zone where the corneal curvature drops off by ≥2D. The energy distribution is based on the maximum corneal steepness (Kmax) value retrieved from the Pentacam HR® tomography: ≤47.0D - 7.2 J/cm2; 47.1-52.0D - 10 J/cm2; ≥52.1D - 15 J/cm2. Thus, the thin protruding areas of the cornea are crosslinked, whereas the parts with a more normal shape are not. The aim is to potentially improve the optical outcome after the treatment.

Patients are randomized to either of the two treatment arms utilizing a computer list of unique random numbers between 1 and 50; an even number will be treated with KXL2 and an uneven number with pCXL. Bilateral inclusion is allowed, and the second eye to be treated will be assigned to the other group, i.e. eye number two will not get the same treatment as eye number 1.

All patients are informed about the procedures and provide oral and written consent before inclusion in the study.

At baseline, before treatment, each eye is evaluated with autorefractometer measurement (Oculus Parc-1®), uncorrected and best spectacle-corrected LogMAR visual acuity, Oculus Pentacam HR® Scheimpflug photography, Oculus CorVis® high-speed Scheimpflug photography, corneal endothelial photography with a specular microscope camera, Goldmann applanation tonometry and biomicroscopy.

For the Pentacam HR® rotating Scheimpflug camera, each eye is photographed using the "25 pictures" program under standardized, mesopic light conditions. Multiple variables will be analyzed, and individual photographs also will be analyzed manually for light backscatter and for the occurrence of a demarcation line, by a masked observer. The corneal biomechanical characteristics are assessed with data from the Oculus CorVis®, and corneal endothelial morphometry, including endothelial cell density is assessed manually and automatically from specular microscopy photographs taken with the Topcon SP-2000 endothelial camera. All investigations are repeated at 1 month, 3 months, 6 months and 12 months after the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients planned for corneal crosslinking.
2. Uni-or bilateral keratoconus diagnosis based on the Amsler-Krumeich grading and the "Total Deviation" keratoconus quantification value from the "Belin-Ambrosio enhanced ectasia" measurements of the Pentacam HR® Scheimpflug camera, and an altered red reflex and/or an irregular cornea seen as distortion of the keratometric mires.
3. Progression of the keratoconus in the eye in question, documented with Scheimpflug photography using the Oculus Pentacam HR® Scheimpflug camera and/or repeated subjective refraction and keratometry.
4. Minimum corneal thickness of 400 μm at the thinnest point after epithelial removal.
5. ≥12 years of age
6. No ocular abnormalities except keratoconus
7. No previous ocular surgery
8. No cognitive insufficiency interfering with the informed consent.

Exclusion Criteria:

1. Age under 12
2. Any corneal abnormalities except keratoconus
3. Previous ocular surgery
4. Cognitive insufficiency

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-03; Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in refraction | 1, 3, 6 and 12 months after the treatment
  Change from baseline in refractive errors, including lower and higher order aberrations in the cornea.

SECONDARY OUTCOMES:
Change from baseline in ETDRS LogMAR visual acuity | 1, 3, 6 and 12 months after the treatment
  Changes from baseline in uncorrected and best spectacle corrected visual acuity assessed with the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol, graded in logarithmic values of the minimal angle of resolution.
Change from baseline in corneal densitometry | 1, 3, 6 and 12 months after the treatment
  Change from baseline in corneal densitometry (corneal light backscatter), assessed with the Oculus Pentacam HR® rotating Scheimpflug camera.
  assessed with the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol, graded in logarithmic values of the minimal angle of resolution.
Change from baseline in corneal biomechanical stability measured with GAT | 1, 3, 6 and 12 months after the treatment
  Change from baseline in biomechanical stability assessed with the Goldmann applanation tonometer (GAT).
Change from baseline in corneal biomechanical stability measured with CorVis® | 1, 3, 6 and 12 months after the treatment
  Change from baseline in biomechanical stability assessed with the Oculus CorVis high-speed Scheimpflug camera.
Change from baseline in corneal endothelial morphometry | 1, 3, 6 and 12 months after the treatment
  Change from baseline in corneal endothelial morphometry, including cell density.

REFERENCES:
- [Derived] Nordstrom M, Schiller M, Fredriksson A, Behndig A. Refractive improvements and safety with topography-guided corneal crosslinking for keratoconus: 1-year results. Br J Ophthalmol. 2017 Jul;101(7):920-925. doi: 10.1136/bjophthalmol-2016-309210. Epub 2016 Nov 29. PMID 27899371